CLINICAL TRIAL: NCT03804476
Title: A Phase 1, Double-Blind, Randomized, Placebo-Controlled, Sequential-Group Study to Assess the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Doses of AER-271 in Healthy Subjects
Brief Title: Phase 1 Study to Assess AER-271
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aeromics, Inc. (Industry)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 174273
Record Dates: First submitted 2019-01-09; First posted 2019-01-15 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Stroke; Stroke, Acute; Stroke, Ischemic
Keywords: stroke; acute ischemic stroke; cerebral edema
MeSH Terms: conditions — Stroke; Ischemic Stroke; Brain Edema | interventions — AER-271

STUDY DESIGN:
Intervention Model Description: A double-blind, randomized, placebo-controlled, sequential-group, single and multiple intravenous dose escalation study conducted in 2 parts. Both Parts A and B will comprise an adaptive design. Part A sentinel dosing will randomize the first 2 subjects 1:1 AER-271:placebo. The remaining 6 subjects in a cohort will be randomized 5:1 AER-271:placebo and administered drug after the Safety Monitoring Board (SMB) has reviewed the first 24 hours of safety data for the first 2 subjects. Part B sentinel dosing will randomize the first 4 subjects 2:2 AER-271:placebo. The remaining 6 subjects in a cohort will be randomized 4:2 AER-271:placebo and administered study drug after the SMB has reviewed the first 24 hours of safety data for the first 4 subjects. Part A will have 6 cohorts and Part B will have 3. Additional cohorts may be enrolled to explore additional dose levels. The planned study design may be modified in accordance with the adaptive features of the clinical study protocol.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The participants, care providers, investigators, outcome assessors, and safety monitoring board will be blind to the administration of AER-271.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AER-271 (Experimental): The experimental drug AER-271 will be administered in this Arm. In Part A single ascending doses will be administered by IV bolus infusion of AER-271 formulated in phosphate buffered normal saline over a 30-min period. In Part B multiple ascending doses of AER-271 will be administered by IV 30-min bolus infusion BID for 72 hours. AER-271 will also be administered as an initial bolus dose over 30-min then continuous infusion over 72 hours.
  Interventions: Drug: AER-271
- Placebo (Placebo Comparator): A placebo control will be administered in this Arm. In Part A phosphate buffered normal saline will be administered over a 30-min period. In Part B multiple doses of phosphate buffered normal saline will be administered by IV 30-min bolus infusion BID for 72 hours. This placebo will also be administered as an initial bolus dose over 30-min then continuous infusion over 72 hours. In both Parts, the volume of placebo administered will be the same as the Experimental Arm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AER-271 — AER-271, the test article for this study.
  Arms: AER-271
Drug: Placebo — Placebo control for this study.
  Arms: Placebo

SUMMARY:
The objective of this Phase 1 trial is to assess the safety, tolerability and pharmacokinetics of AER-271 in health subjects.

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled, sequential-group study to assess the safety, tolerability and pharmacokinetics of single ascending dose and multiple ascending doses of intravenously (IV) administered AER-271 in healthy human subjects. AER-271 is an Aquaporin-4 inhibitor designed to prevent brain swelling in severe ischemic stroke. The study will be conducted in 2 parts: Part A is a single ascending dose, sequential group study. The subsequent Part B is a multiple ascending dose, sequential group study. Both Parts A and B will follow an adaptive design including the use of Sentinel Dosing.

The primary objectives of this study are to assess the safety and tolerability of single and multiple IV doses and continuous infusion of AER-271 in healthy subjects. Secondary objectives include: determining the pharmacokinetics of AER-271 and AER-270 following administration of AER-271, determining the dose proportionality for AER-270 and 271, and comparing the effects of continuous infusion versus multiple bolus doses on AER-271 exposure and adverse events. An additional exploratory objective of this study is to evaluate the effects of AER-271 on electrocardiogram parameters including QT interval corrected for heart rate. Data from this trial will also be used to develop a protocol for a subsequent Phase 2 clinical trial in stroke patients.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, of any ethnic origin, between 18 and 45 years of age, inclusive, at Screening.
2. Body mass index between 18.0 and 32.0 kg/m2, inclusive, at Screening.
3. In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, vital sign measurements, and clinical laboratory evaluations (congenital nonhemolytic hyperbilirubinemia [eg, suspected Gilbert's syndrome, as determined by total bilirubin and indirect bilirubin] is acceptable) at Screening and/or Check-in, as assessed by the Investigator.
4. Male subjects must be surgically sterile for at least 90 days or, for males capable of fathering children who are sexually active with female partners of childbearing potential, will use the required contraception methods, and will refrain from donating sperm from the time of the first dose until 90 days after the final dosing occasion.
5. Female subjects must be:

   * postmenopausal, defined as at least 12 months post cessation of menses (without an alternative medical cause) with a screening serum follicle-stimulating hormone (FSH) level > 40 mIU/mL, or
   * permanently sterile following hysterectomy, Essure procedure, bilateral salpingectomy, bilateral oophorectomy, or confirmed tubal occlusion (not tubal ligation).
6. Venous access sufficient for IV infusions.
7. Able to comprehend and willing to sign an Informed Consent Form (ICF) and to abide by the study restrictions.

Exclusion Criteria:

1. Female subjects who are pregnant or lactating.
2. Have any clinically significant abnormal physical examination finding at Check-in.
3. Have any clinically significant medical history, as determined by the Investigator.
4. History of seizure disorder, even if currently not receiving anticonvulsant medications.
5. Part B only: Have acute suicidality, as evidenced by answering "yes" for Question 4 or Question 5 on the C-SSRS, indicating active suicidal ideation with any intent to act at Screening and Check-in.
6. Part B only: Have a history of suicidal behavior such that a determination of "yes" is made on the Suicidal Behavior section of the C-SSRS for "Actual Attempt," "Interrupted Attempt," "Aborted Attempt," or "Preparatory Acts or Behavior" at Screening and Check-in.
7. History or clinical manifestations of clinically significant metabolic (including diabetes mellitus, hypercholesterolemia, or dyslipidemia), hematologic, pulmonary, cardiovascular, gastrointestinal (cholecystectomy and appendectomy are acceptable), neurologic, hepatic, renal, urologic, immunologic, or psychiatric disorders (a history of mild depression, currently not receiving therapy, is acceptable), as determined by the Investigator.
8. Have any clinically significant allergic condition (excluding non-active hay fever), as determined by the Investigator.
9. Have a significant history of drug allergy, as determined by the Investigator.
10. Have a clinically significant abnormality in oral temperature, respiratory rate, or supine pulse rate or blood pressure at Screening and prior to first dose that, in the opinion of the Investigator, increases the risk of participating in the study.
11. Electrocardiogram findings that meet any of the following criteria at Screening or Day-1 (if out of range, ECG may be repeated twice, and the triplicate average will be used):

    * QTcF >450 msec confirmed by repeat measurement,
    * QRS duration > 120 msec,
    * PR interval >220 msec,
    * findings which would make QTc measurements difficult or QTc data uninterpretable.
12. History of additional risk factors for torsades de pointe (eg, heart failure, hypokalemia, family history of long QT syndrome).
13. Have clinically significant arrhythmias or sinus pauses identified in the continuous 12-lead ECG monitoring on Day -1, as determined by the Investigator.
14. Have any clinically significant abnormal laboratory safety findings at Screening and Check-in, as determined by the Investigator or designee (one repeat assessment is acceptable). Note: Liver function tests (eg, AST, ALT, total bilirubin, GGT) and inflammatory response markers (eg, white blood cell and absolute neutrophil and monocyte counts) must be within the normal range at Screening (one repeat assessment is acceptable) (after Screening this will be as determined by the Investigator).
15. A positive hepatitis virus test (hepatitis B surface antigen or hepatitis C virus antibody) or a positive human immunodeficiency virus antibody test (or p24 antigen) at Screening.
16. Have had a clinically significant illness within 4 weeks of first dose, as determined by the Investigator (or designee).
17. Alcohol consumption of > 21 units per week for males and > 14 units per week for females. Note: One unit of alcohol equals 12 oz (360 mL) beer, 1.5 oz (45 mL) liquor, or 5 oz (150 mL) wine.
18. Significant history of alcoholism or drug/chemical abuse, as determined by the Investigator.
19. An active smoker or user of other forms of tobacco. Former smokers or tobacco users must have refrained from smoking or using other forms of tobacco for at least 6 months prior to dosing on Day 1 until the Follow-up visit.
20. Have donated blood from 90 days prior to Screening, platelets from 42 days prior to Screening, or plasma from 7 days prior to Screening until 56 days after the Follow-up visit.
21. Have received another investigational drug within 30 days prior to randomization.
22. Have received known inhibitors or inducers of CYP1A2 or any medications or herbal remedies, including St. John's Wort, known to chronically alter drug absorption or elimination processes within 30 days prior to first dose administration, until the Follow-up visit, unless in the opinion of the Investigator (or designee), Medical Monitor, and/or Aeromics, the medication will not interfere with the study procedures or compromise safety.
23. Use of any prescription medications/products within 14 days prior to randomization, or use of nonprescription, over-the-counter medication/products, including vitamins, minerals, and phytotherapeutic/herbal/plant-derived preparations, within 7daysprior to randomization until the Follow-up visit. Exceptions may be made by the Medical Monitor, Investigator (or designee), and/or Aeromics on a case-by-case basis. Intermittent use of acetaminophen at moderate daily doses (eg, ≤ 1g per day for ≤2 consecutive days) may be allowed at the discretion of the Investigator.
24. Positive urine drug screen at Screening (not including cotinine or alcohol) or Check-in (including cotinine and alcohol), confirmed by repeat.
25. Consumption of foods and beverages containing poppy seeds, grapefruit, or Seville oranges within 7 days prior to Check-in until the Follow-up visit.
26. Subjects unwilling to refrain from strenuous exercise from 7 days before Check- in until the Follow-up visit.
27. Consumption of alcohol-containing foods and beverages within 72 hours prior to Check-in until the Follow-up visit.
28. Consumption of caffeine-containing foods and beverages within 72 hours prior to Check-in until discharge on Day 3 for Part A or on Day 12 for Part B.
29. Have previously taken part in or withdrawn from this study.
30. Subjects who, in the opinion of the Investigator, should not participate in this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2019-07-18 (Actual); Study Completion 2019-08-28 (Actual)

PRIMARY OUTCOMES:
Number of patients that experience adverse events | Changes from baseline through day 5-7 for Part A and day 15-17 Part B.
  Observation for signs and symptoms of adverse events
Number of patients that experience serious adverse events | Changes from baseline through day 5-7 for Part A and day 15-17 Part B.
  Observation for signs and symptoms of serious adverse events
Number of patients with significant changes in ALT levels | Changes from baseline through day 5-7 for Part A and day 15-17 Part B.
  Patients with serum Alanine Aminotransferase exceeding or below normal values will be reported with the concentration in IU/L
Number of patients with significant changes in AST levels | Changes from baseline through day 5-7 for Part A and day 15-17 Part B.
  Patients with serum Aspartate Aminotransferase exceeding or below normal values will be reported with the concentration in IU/L
Number of patients with significant changes in GGT levels | Changes from baseline through day 5-7 for Part A and day 15-17 Part B.
  Patients with serum Gamma-Glutamyl Transferase exceeding or below normal values will be reported with the concentration in IU/L
Number of patients with significant changes in WBC | Changes from baseline through day 5-7 for Part A and day 15-17 Part B.
  Patients with White Blood Cell Count exceeding or below normal values will be reported in count/uL
Number of patients with significant changes in RBC | Changes from baseline through day 5-7 for Part A and day 15-17 Part B.
  Patients with Red Blood Cell Count exceeding or below normal values will be reported in count/uL
Number of patients with significant changes in Albumin levels | Changes from baseline through day 5-7 for Part A and day 15-17 Part B.
  Patients with serum Albumin exceeding or below normal values will be reported with the concentration in g/dL
Number of patients with significant changes in Bilirubin levels | Changes from baseline through day 5-7 for Part A and day 15-17 Part B.
  Patients with Bilirubin exceeding or below normal values will be reported with the concentration in mg/dL
Number of patients with significant changes in Platelet counts | Changes from baseline through day 5-7 for Part A and day 15-17 Part B.
  Patients with Platelet counts exceeding or below normal values will be reported as count/uL
Number of patients with significant changes in Hematocrit | Changes from baseline through day 5-7 for Part A and day 15-17 Part B.
  Patients with Hematocrit exceeding or below normal values will be reported as a %
Number of patients with significant changes in Creatinine | Changes from baseline through day 5-7 for Part A and day 15-17 Part B.
  Patients with serum Creatinine exceeding or below normal values will be reported with the concentration in mg/dL
Number of patients with significant changes in Alkaline Phosphatase levels | Changes from baseline through day 5-7 for Part A and day 15-17 Part B.
  Patients with serum Alkaline Phosphatase exceeding or below normal values will be reported with the concentration in IU/L
Number of patients with significant changes in Cholesterol levels | Changes from baseline through day 5-7 for Part A and day 15-17 Part B.
  Patients with Cholesterol exceeding or below normal values will be reported with the concentration in mg/dL
Number of patients with significant changes in Respiratory Rate | Changes from baseline through day 5-7 for Part A and day 15-17 Part B.
  Patients with changes in Respiratory Rate will be reported in count/min
Number of patients with significant changes in Pulse Rate | Changes from baseline through day 5-7 for Part A and day 15-17 Part B.
  Patients with changes in Pulse Rate will be reported in count/min
Number of patients with significant changes in Oral Temperature | Changes from baseline through day 5-7 for Part A and day 15-17 Part B.
  Patients with changes in Oral Temperature above normal will be reported in degrees Celcius (C)
Number of patients with significant changes in Blood Pressure | Changes from baseline through day 5-7 for Part A and day 15-17 Part B.
  Patients with changes in Supine Blood Pressure exceeding or below normal values will be reported in mmHg systolic over diastolic
Number of patients exhibiting changes in Physical Examination | Changes from baseline through day 5-7 for Part A and day 15-17 Part B.
  Number of patients exhibiting any changes in the physical examination during this period will be reported.

SECONDARY OUTCOMES:
Pharmacokinetic parameter: Mean Cmax +/- standard deviation | This pharmacokinetic parameter will be assessed at the end of each of 6 cohorts in the SAD study (within 1-2 weeks of final blood sample collection) and 3 cohorts in the MAD study (within 1-2 weeks of final blood sample collection).
  Maximum concentration of AER-271 and AER-270 derived from plasma concentration-time profile (ng/mL)
Pharmacokinetic parameter: Mean AUC +/- standard deviation | This pharmacokinetic parameter will be assessed at the end of each of 6 cohorts in the SAD study (within 1-2 weeks of final blood sample collection) and 3 cohorts in the MAD study (within 1-2 weeks of final blood sample collection).
  Area Under the Curve for AER-271 and AER-270 derived from plasma concentration-time profile (hr*ng/mL)
Pharmacokinetic parameter: Mean CL +/- standard deviation | This pharmacokinetic parameter will be assessed at the end of each of 6 cohorts in the SAD study (within 1-2 weeks of final blood sample collection) and 3 cohorts in the MAD study (within 1-2 weeks of final blood sample collection).
  Clearance of AER-271 derived from plasma concentration-time profile (mL/hr/kg)
Pharmacokinetic parameter: Mean T1/2 +/- standard deviation | This pharmacokinetic parameter will be assessed at the end of each of 6 cohorts in the SAD study (within 1-2 weeks of final blood sample collection) and 3 cohorts in the MAD study (within 1-2 weeks of final blood sample collection).
  Half-life of AER-271 and AER-270 derived from plasma concentration-time profile (hr)
Pharmacokinetic parameter: Mean Vss +/- standard deviation | This pharmacokinetic parameter will be assessed at the end of each of 6 cohorts in the SAD study (within 1-2 weeks of final blood sample collection) and 3 cohorts in the MAD study (within 1-2 weeks of final blood sample collection).
  Steady state volume of distribution of AER-271 derived from plasma concentration-time profile (mL/kg)
Changes in ECG Parameters: Mean QTcF +/- standard deviation | Changes from baseline through day 5-7 for Part A and day 15-17 Part B.
  QT Interval Corrected by Fridericia's Formula (msec)
Changes in ECG Parameters: Mean QRS +/- standard deviation | Changes from baseline through day 5-7 for Part A and day 15-17 Part B.
  QRS Duration (msec)
Changes in ECG Parameters: Mean PR +/- standard deviation | Changes from baseline through day 5-7 for Part A and day 15-17 Part B.
  PR Interval (msec)

CONTACTS AND LOCATIONS:
Overall Officials: Paul R McGuirk, PhD, Principal Investigator — Aeromics, Inc.; Alex King, MD, Principal Investigator — Covance
Locations (1):
- Covance Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No